CLINICAL TRIAL: NCT00298259
Title: Prospective Randomised Trial of Operative Fixation of Fractured Ribs in Patients With Flail Chest
Brief Title: Trial of Operative Fixation of Fractured Ribs in Patients With Flail Chest
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Alfred (Other)
Responsible Party: Principal Investigator, Silvana Marasco, Associate Professor Silvana Marasco, The Alfred
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 50/06
Record Dates: First submitted 2006-03-01; First posted 2006-03-02 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Flail Chest; Ventilation
MeSH Terms: conditions — Flail Chest; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ORIF (Active Comparator): open reduction internal fixation of fractured ribs in flail chest patients
  Interventions: Procedure: operative fixation of fractured ribs
- conservative management (No Intervention): current standard conservative management

INTERVENTIONS:
Procedure: operative fixation of fractured ribs — ORIFof fractured ribs in flail chest patients
  Arms: ORIF

SUMMARY:
Background: Fracture of several ribs in more than one place as the result of trauma, leads to paradoxical movement of the chest wall and ventilatory failure. The mainstay of management in these patients has traditionally been analgesia and positive pressure ventilation to splint the chest wall and allow healing of the ribs to begin. However, this management option leads to prolonged intensive care unit (ICU) stay with increasing complication rates as patients remain on a ventilator for prolonged periods. Patients often remain on a ventilator for two to three weeks while waiting for enough rib healing to provide sufficient chest wall stability to allow the patient to take over all their breathing themselves. Until that time, patients are at risk of pneumonia and sepsis and other complications. Long term disabilities which have been reported in these patients include ongoing pain syndromes, inability to return to work, particularly manual type labour and cosmetic chest wall deformities.

An alternative treatment strategy is to operatively fix the ribs. By fixing the ribs operatively, the patient no longer requires internal pneumatic stabilization (provided by mechanical ventilation) and can be weaned from the ventilator within days rather than weeks. This can potentially lead to earlier discharge from the intensive care unit, and an avoidance of the multiple complications which arise in the ventilated patient. Rib fixation may also lead to less pain and deformity, improved mobility in the post injury phase and earlier return to work.

Hypothesis: that early operative fixation of ribs in patients presenting with flail chest secondary to trauma will result in less mechanical ventilatory requirements, earlier discharge from the intensive care unit and lower rate of complications associated with prolonged mechanical ventilation. This will lead to cost savings in the treatment of these patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with multiple (>3) fractured ribs between the level of ribs 3 to 10 resulting in a paradoxical movement of the chest wall -

Exclusion Criteria:

* age > 75 years
* Spinal injuries which would preclude placement of the patient in a lateral decubitus position
* Open rib fractures with soiling or infection
* Severe head injury
* Uncorrected coagulopathy
* Adult respiratory distress syndrome
* Sepsis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-01; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Mechanical ventilation hours | open
intensive care stay hours | open

CONTACTS AND LOCATIONS:
Overall Officials: Silvana Marasco, FRACS, Principal Investigator — The Alfred
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia